CLINICAL TRIAL: NCT07229157
Title: A Phase 1, Randomized, Double-blind, Placebo- and Positive-controlled, Parallel Group Study With Nested Crossover Comparison to Assess the Effect of Maridebart Cafraglutide on QT/QTc Intervals in Participants Living With Overweight or Obesity
Brief Title: Effect of Maridebart Cafraglutide on the Heart's Electrical Activity
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20250003
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Maridebart Cafraglutide; AMG 133; QT/QTc Intervals
MeSH Terms: conditions — Overweight; Obesity | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): In treatment period 1, participants will receive placebo for moxifloxacin.
  In treatment period 2, participants will receive maridebart cafraglutide.
  In treatment period 3, participants will receive placebo for moxifloxacin.
  Interventions: Drug: Maridebart Cafraglutide; Drug: Placebo for Moxifloxacin
- Group 2A (Experimental): In treatment period 1, participants will receive moxifloxacin.
  In treatment period 2, participants will receive placebo for maridebart cafraglutide.
  In treatment period 3, participants will receive placebo for moxifloxacin.
  Interventions: Drug: Moxifloxacin; Drug: Placebo for Maridebart Cafraglutide; Drug: Placebo for Moxifloxacin
- Group 2B (Experimental): In treatment period 1, participants will receive placebo for moxifloxacin.
  In treatment period 2, participants will receive placebo for maridebart cafraglutide.
  In treatment period 3, participants will receive moxifloxacin.
  Interventions: Drug: Moxifloxacin; Drug: Placebo for Maridebart Cafraglutide; Drug: Placebo for Moxifloxacin

INTERVENTIONS:
Drug: Maridebart Cafraglutide — Participants will receive maridebart cafraglutide SC.
  Other Names: AMG 133
  Arms: Group 1
Drug: Moxifloxacin — Participants will receive moxifloxacin orally.
  Arms: Group 2A; Group 2B
Drug: Placebo for Maridebart Cafraglutide — Participants will receive placebo for maridebart cafraglutide SC.
  Arms: Group 2A; Group 2B
Drug: Placebo for Moxifloxacin — Participants will receive placebo for moxifloxacin orally.

SUMMARY:
The main objective of this trial is to evaluate the effect of maridebart cafraglutide subcutaneously (SC) on the placebo-corrected, change from baseline in QT interval corrected for heart rate using Fridericia's formula in participants living with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria

To take part in the trial, participants must meet all of the following:

1. Provide signed and dated informed consent before any trial procedures.
2. Be able to understand the trial requirements, sign the consent form, and follow trial restrictions.
3. Male or female, of any race, between 18 and 60 years old (inclusive).

   * Females must not be pregnant or breastfeeding.
   * Males and females who could become pregnant must agree to use effective birth control as specified in the protocol.
4. Body mass index (BMI) between 25.0 and 35.0 kg/m^2 (inclusive).
5. No major changes in diet or lifestyle in the past 3 months, based on self-report.
6. Stable body weight (less than 5 kg change) in the past 3 months, based on self-report.
7. Blood potassium, calcium, and magnesium within the normal range at screening and at check-in for the first treatment period.
8. Participants with controlled high blood pressure, cholesterol problems, or hypothyroidism on stable treatment for at least 3 months may be included (except for medicines known to affect heart rhythm or interact with moxifloxacin). Other mild, stable health conditions may be allowed with approval from the investigator and medical monitor.

Exclusion Criteria

Participants will not be able to take part if they meet any of the following:

Medical Conditions

1. Any significant medical condition or abnormal test result that, in the opinion of the investigator, could pose a risk or interfere with trial participation.
2. History of diabetes (any type, except past gestational diabetes), or Haemoglobin A1c (HbA1c) ≥ 6.5% at screening.
3. History of pancreatitis within the past year, or high blood tests suggesting pancreatic problems (lipase/amylase > 2× normal, or fasting triglycerides > 500 mg/dL).
4. Liver enzymes (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) more than 2× the upper limit of normal.
5. Kidney function (estimated glomerular filtration rate [eGFR]) < 70 mL/min/1.73 m^2.
6. Cancer within the last 5 years (except treated nonmelanoma skin cancers or in situ cervical/breast lesions).
7. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2.
8. Uncontrolled thyroid disease (abnormal thyroid-stimulating hormone [TSH] outside 0.4-6.0 mIU/L).
9. Contraindications to moxifloxacin, including history of tendon disorders with quinolone use.
10. History of gastrointestinal surgery or disease that may affect absorption of oral drugs (other than uncomplicated appendectomy or hernia repair).
11. Inability to swallow pills.
12. History of significant esophageal, stomach, or bowel disorders (eg, ulcers, bleeding, Crohn's disease, ulcerative colitis, irritable bowel syndrome, gastroparesis).
13. Current or recent suicidal thoughts (per Columbia Suicide Severity Rating Scale [C-SSRS]).
14. Lifetime history of suicide attempt or behavior.
15. Major depressive disorder within the past 2 years.
16. History of other serious psychiatric disorders (eg, schizophrenia, bipolar disorder).
17. High depression score (patient health questionnaire-9 [PHQ-9] ≥ 15).
18. History or current signs of heart disease (eg, heart attack, congenital defects, valve disease, angina, bypass or stent).
19. History of ischemic optic neuropathy (eye damage from poor blood flow).
20. Diagnosis of sleep apnea. Diagnostic Tests
21. Positive test for human immunodeficiency virus (HIV).
22. Positive test for hepatitis B or C (exceptions apply for prior vaccination or resolved infection).
23. Abnormal vital signs: average blood pressure > 140/90 mmHg or < 90/50 mmHg, or heart rate > 110 or < 40 bpm.
24. Abnormal ECG findings at screening or check-in, including:

    * QTcF > 450 ms (males) or > 470 ms (females).
    * QRS > 120 ms, PR > 220 ms, AV block (2nd or 3rd degree).
    * Findings that make QTc measurement unreliable.
    * Risk factors for dangerous arrhythmias (eg, heart failure, low potassium, long QT syndrome).
    * Clinically significant arrhythmias. Medications
25. Use of drugs that affect absorption, metabolism, or elimination within 30 days of dosing.
26. Use of drugs known to prolong QT/QTc within 30 days of dosing.
27. Use of prescription drugs (other than hormone replacement or contraception) within 14 days of dosing.
28. Use of long-acting/slow-release medicines still active within 14 days of dosing.
29. Use of non-prescription products (vitamins, supplements, herbal products) within 7 days of dosing.
30. Use of glucagon-like peptide-1 (GLP-1) or glucose-dependent insulinotropic polypeptide (GIP) receptor agonists/antagonists within 3 months of check-in.

    Other Clinical Trial Experience
31. Participation in another investigational drug trial within 30 days or 5 drug half-lives (whichever is longer).
32. Previous exposure to maridebart cafraglutide in this or another trial. Lifestyle
33. Alcohol use > 21 units/week (men) or > 14 units/week (women).
34. Alcohol use within 48 hours before check-in.
35. Positive drug screen or alcohol test at screening or check-in.
36. History of alcohol or drug abuse within 1 year.
37. Use of tobacco/nicotine products within 3 months, or positive cotinine test.
38. Use of caffeine within 48 hours of screening or check-in.
39. Consumption of grapefruit, Seville orange, or related products within 7 days of check-in.
40. Consumption of poppy seed-containing foods within 7 days of check-in. Other
41. Receipt of blood products within 2 months before check-in.
42. Blood donation within 3 months; plasma donation within 2 weeks; platelet donation within 6 weeks.
43. Poor veins for blood draws.
44. Any other reason, in the opinion of the investigator, the participant should not take part.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in QTcF for Maridebart Cafraglutide | Up to Day 171
  Change from baseline in QTcF for maridebart cafraglutide will be the dependent variable for calculation of model-derived placebo-corrected, change from baseline in QTcF after maridebart cafraglutide dosing.

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve Over the Dosing Interval (AUCtau) of Maridebart Cafraglutide | Up to Day 171
Maximum Observed Concentration (Cmax) of Maridebart Cafraglutide | Up to Day 171
Change from Baseline in Heart Rate | Up to Day 171
  Change from baseline in heart rate will be used as the dependent variable for calculation of model-derived placebo-corrected, change from baseline in HR for the by-time point analysis.
Change from Baseline in PR Interval | Up to Day 171
  Change from baseline in PR Interval will be used as the dependent variable for calculation of model-derived placebo-corrected, change from baseline in PR for the by-time point analysis.
Change from Baseline in QRS Duration | Up to Day 171
  Change from baseline in QRS Duration will be used as the dependent variable for calculation of model-derived placebo-corrected, change from baseline in QRS for the by-time point analysis.
Categorical Outliers for QTcF | Up to Day 171
Categorical Outliers for HR | Up to Day 171
Categorical Outliers for PR | Up to Day 171
Categorical Outliers for QRS | Up to Day 171
Number of Participants with Treatment-emergent Changes in Electrocardiogram (ECG) Morphology | Up to Day 171
Change from Baseline in QTcF for Moxifloxacin | Up to Day 171
  Change from baseline in QTcF for moxifloxacin will be used as the dependent variable for calculation of model-derived placebo-corrected, change from baseline in QTcF after moxifloxacin dosing for both the assay sensitivity and by-time point analysis.
Number of Participants with Treatment-emergent Adverse Events and Serious Adverse Events | Up to Day 232
Number of Participants with Anti-maridebart Cafraglutide Antibody Formation | Up to Day 232

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Fortrea Clinical Research Unit - Daytona Beach, Daytona Beach, Florida
  - Fortrea Clinical Research Unit - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com